CLINICAL TRIAL: NCT06101511
Title: Driving Pressure During General Anesthesia for Minimally Invasive Abdominal Surgery (GENERATOR) - a Randomized Clinical Trial
Brief Title: Driving Pressure During General Anesthesia for Minimally Invasive Abdominal Surgery (GENERATOR)
Acronym: GENERATOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other); HagaZiekenhuis (Other); Dijklander Ziekenhuis (Other); The Netherlands Cancer Institute (Other); Isala (Other); Maasstad Hospital (Other); Medisch Spectrum Twente (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Hospital Universitario La Fe (Other); Ospedale Policlinico San Martino (Other); University Hospital Carl Gustav Carus (Other); Medical University Innsbruck (Other); Spaarne Gasthuis (Other); Zaans Medical Center (Unknown); Alrijne Hospital (Other); Albert Schweitzer Hospital (Other); Maastricht University Medical Center (Other); Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Professor of Intensive Care Medicine, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL82971.018.23
Record Dates: First submitted 2023-07-19; First posted 2023-10-26 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Complications; Surgery
Keywords: Minimally invasive abdominal surgery; Mechanical ventilation; Positive end-expiratory pressure; Driving pressure; Postoperative pulmonary complications; Recruitment maneuver
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized high PEEP strategy with recruitment maneuvers (Experimental): The intervention is intraoperative ventilation using the available ventilator with individualized high positive end-expiratory pressure (PEEP) titrated to the lowest driving pressure (ΔP) with recruitment maneuvers (RMs). After abdominal insufflation, patients randomized to the individualized high PEEP with RMs group will receive a RM followed by a 'decremental PEEP trial'. This is followed by a second RM after which PEEP is set at the level indicated by the decremental PEEP trial.
  Interventions: Procedure: Intraoperative ventilation with individualized high PEEP titrated to the lowest ΔP with RMs
- Standard low PEEP strategy without recruitment maneuvers (No Intervention): Patients randomized to the standard low PEEP group will receive 5 cm H2O PEEP for the complete duration of general anesthesia. They will neither receive one of the planned RMs nor a decremental PEEP trial.

INTERVENTIONS:
Procedure: Intraoperative ventilation with individualized high PEEP titrated to the lowest ΔP with RMs — The intervention is intraoperative ventilation using the available ventilator with individualized high PEEP titrated to the lowest ΔP with RMs. After abdominal insufflation, patients randomized to the individualized high PEEP with RMs group will receive a RM followed by a 'decremental PEEP trial'. This is followed by a second RM after which PEEP is set at the level indicated by the decremental PEEP trial
  Other Names: Individualized high PEEP strategy with recruitment maneuvers
  Arms: Individualized high PEEP strategy with recruitment maneuvers

SUMMARY:
The purpose of this international multicenter, patient and outcome-assessor blinded randomized controlled trial is to determine whether the application of an individualized high Positive End Expiratory Pressure (PEEP) strategy with recruitment maneuvers, aiming at avoiding an increase in the driving pressure during intraoperative ventilation, protects against the development of postoperative pulmonary complications in patients undergoing minimally invasive abdominal surgery.

ELIGIBILITY:
Inclusion criteria:

1. age > 18 years; AND
2. scheduled for minimally invasive abdominal surgery; AND
3. at increased (i.e., intermediate or high) risk of PPCs according to the 'Assess Respiratory risk in Surgical Patients in Catalonia' (ARISCAT) risk score (≥ 26 points, see Appendix I); OR at increased risk of PPCs based on the combination of age > 40 years, scheduled surgery lasting > 2 hours and planned to receive an intra-arterial catheter for blood pressure monitoring during the surgery; AND
4. signed written informed consent

Exclusion criteria:

1. planned for open abdominal surgery;
2. planned for surgery in lateral or prone position;
3. planned for combined abdominal and intra-thoracic surgery
4. confirmed pregnancy;
5. consent for another interventional trial during anesthesia;
6. having received invasive ventilation > 30 minutes within the last five days;
7. any previous lung surgery;
8. history of previous severe chronic obstructive pulmonary disease (COPD) with (noninvasive) ventilation or oxygen therapy at home or repeated systemic corticosteroid therapy for acute exacerbations of COPD;
9. history of acute respiratory distress syndrome (ARDS);
10. expected to require postoperative ventilation;
11. expected hemodynamic instability or intractable shock;
12. severe cardiac disease (New York Heart Association class III or IV, acute coronary syndrome or persistent ventricular tachyarrhythmia's).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1806 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants developing one or more postoperative pulmonary complications (PPCs) | The first 5 postoperative days
  A composite of the following pulmonary complications: mild respiratory failure; severe respiratory failure; bronchospasm; suspected pulmonary infection; pulmonary infiltrate; aspiration pneumonitis; atelectasis; acute respiratory distress syndrome (ARDS); pleural effusion; cardiopulmonary edema; pneumothorax

SECONDARY OUTCOMES:
Intraoperative complications | For the duration of general anesthesia, these outcomes are scored every hour up to a maximum of 18 hours
  Including: any episode of desaturation; any episode of hypotension; any need for vasoactive agents, either as bolus or continuous administration, defined as more than needed to compensate for vasodilating effects of anesthesia as judged by the attending anesthesiologist and any new arrhythmias needing intervention
Intraoperative fluid strategy | During general anesthesia
  Including the total amount of fluids administered during anesthesia, including the amounts of colloids, crystalloids, and blood products
Impaired wound healing | The first 5 postoperative days
  Impaired wound healing, as judged and mentioned in the medical record by the attending ward physician;
Postoperative extrapulmonary complications | The first 5 postoperative days
  Including: sepsis; septic shock; extrapulmonary infection; anastomotic leak and acute renal failure
Mortality | Postoperative day 5, day 30 and day 90
  All-cause mortality at day 5, day 30 and 90, and in-hospital mortality
Length of stay | Postoperatively until the end of the 90 day follow-up period
  Length of hospital stay (days); length of ICU admission if applicable (days);
Oxygen use | The first 5 postoperative days
  Postoperative supplemental oxygen use (days). Presence, duration and levels of postoperative supplemental oxygen
Antibiotics use | The first 5 postoperative days
  Use of antibiotics for pneumonia (proportion of patients who received antibiotics)
Thoracic imaging | The first 5 postoperative days
  Occurence of imaging (chest X-ray, computed tomography scan). Proportion of patients who underwent thoracic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Schultz, Professor, Study Chair — Amsterdam University Medical Center, location AMC; Markus Hollmann, Professor, Principal Investigator — Amsterdam University Medical Center, location AMC; David van Meenen, PhD, Principal Investigator — Amsterdam University Medical Center, location AMC; Sabrine Hemmes, PhD, Principal Investigator — Amsterdam University Medical Center, location AMC
Locations (1):
- Amsterdam University Medical Center, Amsterdam, Noordholland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers can contact the Principal Investigator for a collaboration after which an agreement will be discussed.
Supporting Information: Study Protocol
Time Frame: After the main paper has been published. No end-date has been specified for now.
Access Criteria: The applicable researcher can contact the Principal investigator with their idea of using the data, preferably accompanied by a statistical analysis plan

REFERENCES:
- [Derived] GENERATOR-investigators. Driving pressure during general anesthesia for minimally invasive abdominal surgery (GENERATOR)-study protocol of a randomized clinical trial. Trials. 2024 Oct 26;25(1):719. doi: 10.1186/s13063-024-08479-x. PMID 39456048